CLINICAL TRIAL: NCT05209932
Title: Development and Evaluation of an Internet Based Adaptation of the New Beginnings Program for Divorced Parents
Brief Title: An Internet Based Adaptation of a Divorce Intervention Beginnings Program for Divorced Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Family Transitions: Programs that Work (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R44HD082967 (NIH)
Record Dates: First submitted 2021-12-19; First posted 2022-01-27 (Actual); Results first posted 2023-01-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-12

CONDITIONS: Divorce
Keywords: divorce; intervention; positive child outcomes

STUDY DESIGN:
Intervention Model Description: Participants were randomized to receive an online parenting program for divorced and separated parents (N=81) or a wait list control condition (N=50)
Who Masked: Investigator
Masking Description: Investigators were not aware of whether the participants were assigned to eNBP or the wait-list control condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online New Beginnings Program (eNBP) (Experimental): The eNBP is a five-hour, asynchronous, fully web-based adaptation of the group NBP. Separate versions for fathers and mothers consist of the same didactic content and interactive exercises, with gender appropriate references, testimonials and video skills demonstrations. Units are highly interactive. Sessions began with a check-in in which parents responded to questions about use of the program skills and were provided with ways to address the challenges they experienced. The skill was then taught using modeling videos, interactive exercises, and testimonials from prior participants. The program then prompted parents to set times to use the skill, identify barriers to using it and select strategies to reduce these barriers. Parents were provided with tip sheets to address challenges in using the skill, downloadable sheets to record use of and competence in using the skill and a downloadable handbook that summarized what was covered in the unit.
  Interventions: Behavioral: Online New Beginnings Program (eNBP)
- wait-list control condition (No Intervention): Parents in the waitlist-control condition were told that they would have access to the eNBP 12 weeks after they completed the pre-test. Twelve weeks after assignment to condition, parents and children were sent links to the posttest

INTERVENTIONS:
Behavioral: Online New Beginnings Program (eNBP) — The eNBP is a five-hour, asynchronous, fully web-based adaptation of the group-based NBP that can be used on a smart phone, tablet or computer. Separate versions for fathers and mothers consist of the same didactic content and interactive exercises, with gender appropriate references, testimonials and video skills demonstrations.
  Arms: Online New Beginnings Program (eNBP)

SUMMARY:
This study is a two-armed randomized controlled trial of the eNew Beginnings Program (eNBP)'s effects on children's mental health problems as well as interparental conflict, parent-child relationship quality and effective discipline. The eNBP is an asynchronous, fully web-based program that was based on the in-person, group NBP, which has been found to strengthen parent-child relationship quality and effective discipline and reduce children's mental health problems in three randomized controlled trials of the NBP involving over 1,800 children. The investigators hypothesized that parents in the eNBP intervention condition would have less interparental conflict and higher parent-child relationship quality and effective discipline than those in the wait-list control condition. The investigators also expected the children whose parents were in the eNBP intervention condition would have fewer internalizing problems and externalizing problems and higher prosocial skills than those with parents in the wait-list control.

DETAILED DESCRIPTION:
This study is a two-armed intervention randomized controlled trial of the eNew Beginnings Program (eNBP)'s effects on children's mental health problems as well as interparental conflict, parent-child relationship quality and effective discipline. The eNBP is an asynchronous, fully web-based program that was based on the in-person, group-based NBP. Three randomized controlled trials of the NBP involving over 1,800 children found positive effects to strengthen parent-child relationship quality and effective discipline and reduce children's mental health problems. The eNBP teaches all the skills in the 10-session NBP. The investigators hypothesized that parents in the eNBP would have less interparental conflict and higher parent-child relationship quality and effective discipline than those in the wait-list control condition following the intervention. The investigators also expected the children whose parents were in the eNBP would have fewer internalizing problems and externalizing problems and higher prosocial skills than those with parents in the wait-list control following the intervention.

Parents and their offspring were recruited using Qualtrics, a leading-edge sample acquisition technology that partners with 20 online panel providers and recruits nationally. Initial sampling criteria were parent was divorced, separated but never married, divorcing, or separating; had one or more children aged 6 to 18; and spoke English. Parents who met these criteria were sent an email with information about the study and a web-based survey that assessed contact with child/ren, access to a computer with high-speed internet or a smart phone and demographics. Interested parents were provided additional information about the study and screened for eligibility by phone. To be eligible, parents had to be divorced, separated but never married, divorcing or separating; have one or more child between 6 and 18; be English speaking; spend at least three hours/week or at least one overnight every other week with their child(ren); and have access to a computer with high-speed internet or a smart phone. The sample consisted of 131 parents randomized to eNBP (N = 81) or wait-list condition (N = 50) and 102 of their adolescent offspring.

Primary outcome measures were measures of interparental conflict, parent-child relationship quality, effective discipline and children's internalizing and externalizing problems and prosocial behavior.

ELIGIBILITY:
Inclusion Criteria:

* Parents divorced, divorcing or separated
* Parents separated but never married
* One or more children aged 6 to 18
* Parents spoke English
* Parents spend at least 3 hours a week with children or have one overnight every other week with their children
* Parents have access to a computer with high speed internet access of a smart phone

Exclusion Criteria:

* Parents who do not meet all of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2020-02-15 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irwin N Sandler, PhD, Principal Investigator — Family Transitions Programs that Work LLC
Locations (1):
- Family Transitions- Programs that Work, LLC, Mesa, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Data Sharing Plan Results from research conducted under this project will be shared in several ways. Manuscripts will be submitted for publication in high-quality peer-reviewed journals, following the NIH Public Access Policy guidelines. Findings will be presented at relevant national conferences for groups such as Association of Family Courts and Conciliators (AFCC), and Society for Prevention Research (SPR).
  We will also share the deidentified data with other researchers when requested.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: January 2022 - no end date
Access Criteria: Contact Study Co-I/PD - Dr. Michele Porter at m.marie.porter@gmail.com Or through the contact us on the company website.
URL: http://www.familytransitions-ptw.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parents were recruited using Qualtrics, a leading-edge sample acquisition technology. To be eligible, parents had to be divorced, separated but never married, divorcing or separating, have one or more child between six and eighteen, speak English, spend at least three hours a week or at least one overnight every other week with their child(ren), and have access to a computer or a smart phone.
  Recruitment and assessment period was from Feb. 15, 2020 through August 31, 2021.
Pre-assignment Details: Participants were randomly assigned to groups after completing an online pre-test assessment.
Groups:
- Wait-list Control Condition: Parents in the waitlist-control condition were told that they would have access to the eNBP 15 weeks after they completed the pre-test. Fifteen weeks after assignment to condition, parents and children were sent links to the posttest
Period: Overall Study
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Started | 140 (Study participation began February 15th for both treatment group and waitlist control. We had rolling treatment groups and rolling control groups (each Friday for 4 weeks we started a new group). We then put off starting any more cohorts late March (2020) when COVID started getting bad. We did rolling posttests too for each cohort. The waitlist control groups were given access to the program approx. 15 weeks after their cohort started. We finished data collection August 31, 2021.) | 93 (Study participation began February 15th for both treatment group and waitlist control. We had rolling treatment groups and rolling control groups (each Friday for 4 weeks we started a new group). We delayed starting new cohorts when COVID started getting bad. We did rolling posttests too for each cohort. The waitlist control groups were given access to the program approx. 15 weeks after their cohort started. Data collection completed August 31, 2021.)
Completed All or Partial Units | 57 (Completed 10 units - 42.0% (N=34) Completed 5-9 units - 8.6% (N=7) Completed 1-4 units- 19.8% (N=16) Completed 0 units - 29.6% (N=24)) | 93 (Completed 10 units- NA Completed 5-9 units -NA Completed 1-4 units- NA Completed 0 units - NA)
Completed | 140 (N= 81 parents and N=59 children) | 93 (N = 50 parents and N = 43 children)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline population in eNBP of 140 participants includes 81 parents and 59 children within the same family who reported data on different measures. The 93 participants in the Wait List control included 50 parents and 43 children within the same family who reported data on different measures.
  140 in eNBP arm includes 81 parent reports and 59 child reports; 93 in Wait list arm includes 50 parent reports and 43 child reports.
Units Other Than Participants: Parent & child report of child/family
Groups:
- eNBP: The sample consisted of 81 parents who reported on 81 children who were randomly assigned and 59 children in these families who provided self report dates.
- Wait List Controls: 50 parents who reported on 50 children in randomly assigned families and 43 children who self-reported in these families.
- Total: Total of all reporting groups
Arm/Group | eNBP | Wait List Controls | Total
Number analyzed (Participants) | 140 | 93 | 233
Number analyzed (Parent & child report of child/family) | 140 | 93 | 233
Age, Continuous [Mean (Standard Deviation); unit: years] — Child age reported by the parents. Parents reported age on one randomly selected index child per family. Population: The unit of analysis (participants) reflects the number of children who were assessed in the participating families in the eNBP (N = 81) and Wait list control (N = 50) conditions. Parents reported age on one randomly selected index child per family.
  years
    number analyzed (Participants) | 81 | 50 | 131
    (all) | 11.56 (3.80) | 13.67 (3.36) | 12.35 (3.77)
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Measure Analysis Population Description: The unit of analysis (participants) reflects the age of parents who were assessed in the participating families in the eNBP (N = 81) and Wait list control (N = 50) conditions
  years
    number analyzed (Participants) | 81 | 50 | 131
    Age of Parent Participant | 40.47 (7.89) | 40.65 (7.62) | 40.54 (7.75)
Sex: Female, Male [Count of Participants; unit: Participants] — Child gender reported by parents. Parents reported sex on one randomly selected index child per family. Population: Gender information for the target child across 131 families was reported by the parents.
  Participants
    number analyzed (Participants) | 81 | 50 | 131
    Gender of Child Participants: Female | 36 | 26 | 62
    Gender of Child Participants: Male | 45 | 24 | 69
    Gender of Parent Participants: Female | 50 | 33 | 83
    Gender of Parent Participants: Male | 31 | 17 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Parent ethnicity reported by parent (child ethnicity question was not collected). Population: Parent ethnicity information by parent report (child ethnicity info was not collected).
  Participants
    number analyzed (Participants) | 81 | 50 | 131
    Hispanic or Latino | 6 | 4 | 10
    Not Hispanic or Latino | 73 | 46 | 119
    Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Parent race reported by parents (child race information was not collected). Population: Parent race information by parent report (child ethnicity info was not collected).
  Participants
    number analyzed (Participants) | 81 | 50 | 131
    American Indian or Alaska Native | 1 | 1 | 2
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 12 | 5 | 17
    White | 64 | 42 | 106
    More than one race | 1 | 2 | 3
    Unknown or Not Reported | 2 | 0 | 2
Children's Perception of Interparental Conflict Scale (Grych et al., 1992) -- Children Report Versio [Mean (Standard Deviation); unit: units on a scale] — Population: Although 102 children between ages 11 and 18 participated in the baseline assessment, only 85 had enough data for their scores on this measure to be included.
  units on a scale
    number analyzed (Participants) | 50 | 35 | 85
    (all) | 1.55 (0.42) | 1.63 (0.09) | 1.58 (0.47)
Children's Perception of Interparental Conflict Scale (Grych et al., 1992) -- Parent Report Version [Mean (Standard Deviation); unit: units on a scale] — Population: Although 131 parents participated in the baseline assessment, only 124 had enough data for their scores on this measure to be included.
  units on a scale
    number analyzed (Participants) | 76 | 48 | 124
    (all) | 1.41 (0.41) | 1.44 (0.47) | 1.42 (0.43)
Children's Report of Parent Behavior Inventory--Acceptance Subscale (Shaefer, 1965)--Parent Report [Mean (Standard Deviation); unit: units on a scale] — Population: Measure Analysis Population Description: Although 131 parents participated in the baseline assessment, only 119 had enough data for their scores on this measure to be included.
  units on a scale
    number analyzed (Participants) | 72 | 47 | 119
    (all) | 4.58 (0.37) | 4.42 (0.55) | 4.52 (0.45)
Children's Report of Parent Behavior Inventory--Acceptance Subscale (Shaefer, 1965)--Child Report [Mean (Standard Deviation); unit: units on a scale] — Population: Although 102 children between ages 11 and 18 participated in the baseline assessment, only 99 had enough data for their scores on this measure to be included.
  units on a scale
    number analyzed (Participants) | 57 | 42 | 99
    (all) | 4.27 (0.65) | 4.17 (0.65) | 4.23 (0.65)
Children's Report of Parent Behavior Inventory--Rejection Subscale (Shaefer, 1965)--Parent Report [Mean (Standard Deviation); unit: units on a scale] — Population: Although 131 parents participated in the baseline assessment, only 123 had enough data for their scores on this measure to be included.
  units on a scale
    number analyzed (Participants) | 75 | 48 | 123
    (all) | 1.44 (0.40) | 1.63 (0.56) | 1.52 (0.48)
Children's Report of Parent Behavior Inventory--Rejection Subscale (Shaefer, 1965)--Child Report [Mean (Standard Deviation); unit: units on a scale] — Population: Although 102 children between ages 11 and 18 participated in the baseline assessment, only 101 had enough data for their scores on this measure to be included.
  units on a scale
    number analyzed (Participants) | 59 | 42 | 101
    (all) | 1.61 (0.48) | 1.71 (0.61) | 1.65 (0.54)
Children's Report of Parent Behavior Inventory-Consistent Discipline (Shaefer, 1965) --Parent Report [Mean (Standard Deviation); unit: units on a scale] — Population: Although 131 parents participated in the baseline assessment, only 122 had enough data for their scores on this measure to be included.
  units on a scale
    number analyzed (Participants) | 74 | 48 | 122
    (all) | 4.63 (0.56) | 4.45 (0.61) | 4.56 (0.58)
Children's Report of Parent Behavior Inventory-Consistent Discipline (Shaefer, 1965) --Child Report [Mean (Standard Deviation); unit: units on a scale] — Population: Although 102 children between ages 11 and 18 participated in the baseline assessment, only 96 had enough data for their scores on this measure to be included.
  units on a scale
    number analyzed (Participants) | 57 | 39 | 96
    (all) | 4.31 (0.73) | 4.17 (0.92) | 4.25 (0.81)
Oregon Discipline Scale - Follow-Through (Oregon Social Learning Center, 1991) -- Parent Report [Mean (Standard Deviation); unit: units on a scale] — Population: Although 131 parents participated in the baseline assessment, only 125 had enough data for their scores on this measure to be included.
  units on a scale
    number analyzed (Participants) | 79 | 46 | 125
    (all) | 3.79 (0.66) | 3.77 (0.64) | 3.78 (0.65)
Oregon Discipline Scale - Follow-Through (Oregon Social Learning Center, 1991) -- Child Report [Mean (Standard Deviation); unit: units on a scale] — Population: Although 102 children between ages 11 and 18 participated in the baseline assessment, only 94 had enough data for their scores on this measure to be included.
  units on a scale
    number analyzed (Participants) | 53 | 41 | 94
    (all) | 3.80 (0.70) | 3.74 (0.66) | 3.77 (0.68)
Child Monitoring Scale (Hetherington et al., 1992) -- Parent Report [Mean (Standard Deviation); unit: units on a scale] — Population: Although 131 parents participated in the baseline assessment, only 124 had enough data for their scores on this measure to be included.
  units on a scale
    number analyzed (Participants) | 77 | 47 | 124
    (all) | 4.44 (0.58) | 4.37 (0.69) | 4.41 (0.63)
Child Monitoring Scale (Hetherington et al., 1992) -- Child Report [Mean (Standard Deviation); unit: units on a scale] — Population: Although 102 children between ages 11 and 18 participated in the baseline assessment, only 93 had enough data for their scores on this measure to be included.
  units on a scale
    number analyzed (Participants) | 55 | 38 | 93
    (all) | 4.11 (0.71) | 4.12 (0.76) | 4.11 (0.73)
Parent Adolescent Communication Scale (Barnes & Olson, 1985) -- Parent Report [Mean (Standard Deviation); unit: units on a scale] — Population: Although 131 parents participated in the baseline assessment, only 130 had enough data for their scores on this measure to be included.
  units on a scale
    number analyzed (Participants) | 80 | 50 | 130
    (all) | 4.42 (0.56) | 4.40 (0.53) | 4.41 (0.54)
Caught in the Middle Scale (Buchanan et al., 1991) -- Child Report [Mean (Standard Deviation); unit: units on a scale] — Population: Although 102 children between ages 11 and 18 participated in the baseline assessment, only 92 had enough data for their scores on this measure to be included.
  units on a scale
    number analyzed (Participants) | 56 | 36 | 92
    (all) | 1.78 (0.69) | 1.89 (0.69) | 1.82 (0.69)
Brief Problem Monitor -- Externalizing Subscale (Achenbach et al., 2011) -- Parent Report [Mean (Standard Deviation); unit: T-score on a scale] — The sum score of the items (range 0-2 for each item) for each individual is converted to T-score, using the algorithm purchased from ASEBA (Achenbach System of Empirically Based Assessment). The range of the T-scores is: 0 (minimum) to 100 (maximum). score of 50 = the fiftieth percentile of normative sample (Achenbach & Rescola, 2001). T-scores of 65 and above are considered sufficiently elevated to be of concern.
  The values shown are the T-score values for the sample. The norms are based on a US national sample. Population: Although 131 parents participated in the baseline assessment, only 126 had enough data for their scores on this measure to be included.
  T-score on a scale
    number analyzed (Participants) | 79 | 47 | 126
    (all) | 54.17 (5.69) | 54.74 (6.77) | 54.39 (6.10)
Brief Problem Monitor -- Externalizing Subscale (Achenbach et al., 2011) -- Child Report [Mean (Standard Deviation); unit: T-score on a scale] — The sum score of the items (range 0-2 for each item) for each individual is converted to T-score, using the algorithm purchased from ASEBA (Achenbach System of Empirically Based Assessment). The range of the T-scores is: 0 (minimum) to 100 (maximum). score of 50 = the fiftieth percentile of normative sample (Achenbach & Rescola, 2001). T-scores of 65 and above are considered sufficiently elevated to be of concern.
  The values shown are the T-score values for the sample. The norms are based on a US national sample. Population: Although 102 children between ages 11 and 18 participated in the baseline assessment, only 97 had enough data for their scores on this measure to be included.
  T-score on a scale
    number analyzed (Participants) | 55 | 42 | 97
    (all) | 54.40 (6.68) | 56.33 (7.80) | 55.23 (7.21)
Brief Problem Monitor -- Internalizing Subscale (Achenbach et al., 2011) -- Parent Report [Mean (Standard Deviation); unit: T-score on a scale] — The sum score of the items (range 0-2 for each item) for each individual is converted to T-score, using the algorithm purchased from ASEBA (Achenbach System of Empirically Based Assessment). The range of the T-scores is: 0 (minimum) to 100 (maximum). score of 50 = the fiftieth percentile of normative sample (Achenbach & Rescola, 2001). T-scores of 65 and above are considered sufficiently elevated to be of concern.
  The values shown are the T-score values for the sample. The norms are based on a US national sample. Population: Although 131 parents participated in the baseline assessment, only 123 had enough data for their scores on this measure to be included.
  T-score on a scale
    number analyzed (Participants) | 79 | 44 | 123
    (all) | 57.27 (6.39) | 57.91 (7.20) | 57.50 (6.67)
Brief Problem Monitor -- Externalizing Subscale (Achenbach et al., 2011) -- Child Report [Mean (Standard Deviation); unit: T-score on a scale] — The sum score of the items (range 0-2 for each item) for each individual is converted to T-score, using the algorithm purchased from ASEBA (Achenbach System of Empirically Based Assessment). The range of the T-scores is: 0 (minimum) to 100 (maximum). score of 50 = the fiftieth percentile of normative sample (Achenbach & Rescola, 2001). T-scores of 65 and above are considered sufficiently elevated to be of concern.
  The values shown are the T-score values for the sample. The norms are based on a US national sample. Population: Although 102 children between ages 11 and 18 participated in the baseline assessment, only 94 had enough data for their scores on this measure to be included.
  T-score on a scale
    number analyzed (Participants) | 54 | 40 | 94
    (all) | 57.74 (7.72) | 58.25 (8.07) | 57.96 (7.83)
Strengths and Difficulties Questionnaire -- Prosocial Subscale (Goodman, 2001) -- Parent Report [Mean (Standard Deviation); unit: Mean item score on a scale] — Each of the 5 items is scored 0-2. The score reported is the mean item score. A high score is a better outcome. Population: Although 131 parents participated in the baseline assessment, only 129 had enough data for their scores on this measure to be included.
  Mean item score on a scale
    number analyzed (Participants) | 81 | 48 | 129
    (all) | 1.65 (0.39) | 1.62 (0.41) | 1.64 (0.40)
Strengths and Difficulties Questionnaire -- Prosocial Subscale (Goodman, 2001) -- Child Report [Mean (Standard Deviation); unit: Mean item score on a scale] — Each of the 5 items is scored 0-2 (range 0-10). The score reported is the mean total score. A higher score is a better outcome. Population: Although 102 children between ages 11 and 18 participated in the baseline assessment, only 101 had enough data for their scores on this measure to be included.
  Mean item score on a scale
    number analyzed (Participants) | 59 | 42 | 101
    (all) | 8.88 (1.31) | 8.33 (1.79) | 8.65 (1.55)

OUTCOME MEASURES:

1. Primary Outcome: Children's Perception of Interparental Conflict Scale (Grych et al., 1992) -- Children Report Version
Description: 15-item scale assessing frequency and intensity of interparental conflict as reported by children. Minimum score = 1; Maximum score = 3. High score is worse outcome
Time Frame: 1 month
Population: Only children between ages 10 and 18 who were interested and whose parents gave permission completed the assessments (N=102).
Measure: Least Squares Mean (Standard Error); unit: Score on the scale
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Number analyzed (Participants) | 59 | 43
Score on the scale | 1.30 (0.04) | 1.47 (0.06)
Statistical Analysis 1: Comparison: Online New Beginnings Program (eNBP) vs Wait-list Control Condition; Test type: Equivalence — Testing the equivalence of the means using two-tailed test; p = 0.02, ANCOVA; Mean Difference (Net) = -0.17, Standard Error of Mean 0.07

2. Primary Outcome: Children's Perception of Interparental Conflict Scale (Grych et al., 1992) -- Parent Report Version
Description: 15-item scale assessing frequency and intensity of interparental conflict as reported by parents. Minimum score = 1; Maximum score = 3. High score is worse outcome
Time Frame: One month
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Number analyzed (Participants) | 81 | 50
score on a scale | 1.15 (0.10) | 1.26 (0.11)
Statistical Analysis 1: Comparison: Online New Beginnings Program (eNBP) vs Wait-list Control Condition; Test type: Equivalence — Testing the equivalence of the means using two-tailed test; p = 0.05, ANCOVA; Mean Difference (Net) = -.11, Standard Error of Mean 0.06

3. Primary Outcome: Children's Report of Parent Behavior Inventory -- Acceptance Subscale (Shaefer, 1965) -- Parent Report Version
Description: 16-item scales to assess parental acceptance completed by parents. Minimum score = 1. Maximum score = 5. High score is better outcome.
Time Frame: 1 month
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Number analyzed (Participants) | 81 | 50
score on a scale | 4.67 (0.11) | 4.54 (0.14)
Statistical Analysis 1: Comparison: Online New Beginnings Program (eNBP) vs Wait-list Control Condition; Test type: Equivalence — Testing the equivalence of the means using two-tailed test; p = 0.07, ANCOVA; Mean Difference (Net) = .13, Standard Error of Mean .07

4. Primary Outcome: Children's Report of Parent Behavior Inventory -- Acceptance Subscale (Shaefer, 1965) -- Child Report Version
Description: 16-item scales to assess parental acceptance completed by children. Minimum score = 1. Maximum score = 5. High score is better outcome.
Time Frame: 1 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Number analyzed (Participants) | 59 | 43
score on a scale | 4.45 (0.06) | 4.29 (0.11)
Statistical Analysis 1: Comparison: Online New Beginnings Program (eNBP) vs Wait-list Control Condition; Test type: Equivalence — Testing the equivalence of the means using two-tailed test; p = 0.17, ANCOVA; Mean Difference (Net) = 0.17, Standard Error of Mean 0.12

5. Primary Outcome: Children's Report of Parent Behavior Inventory -- Rejection Subscale (Shaefer, 1965) -- Parent Report Version
Description: 16-item scales to assess parental rejection completed by parents. Minimum score = 1. Maximum score = 5. High score is worse outcome.
Time Frame: 1 month
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Number analyzed (Participants) | 81 | 50
score on a scale | 1.41 (0.11) | 1.63 (0.14)
Statistical Analysis 1: Comparison: Online New Beginnings Program (eNBP) vs Wait-list Control Condition; Test type: Equivalence — Testing the equivalence of the means using two-tailed test; p = 0.002, ANCOVA; Mean Difference (Final Values) = -0.22, Standard Error of Mean 0.07

6. Primary Outcome: Children's Report of Parent Behavior Inventory -- Rejection Subscale (Shaefer, 1965) -- Child Report Version
Description: 16-item scales to assess parental rejection completed by children. Minimum score = 1. Maximum score = 5. High score is worse outcome.
Time Frame: 1 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Number analyzed (Participants) | 59 | 43
score on a scale | 1.40 (0.05) | 1.62 (0.09)
Statistical Analysis 1: Comparison: Online New Beginnings Program (eNBP) vs Wait-list Control Condition; Test type: Equivalence — Testing the equivalence of the means using two-tailed test; p = 0.03, ANCOVA; Mean Difference (Net) = -0.22, Standard Error of Mean 0.10

7. Primary Outcome: Children's Report of Parent Behavior Inventory -- Consistency Discipline Subscale (Shaefer, 1965) -- Parent Report Version
Description: 8-item scales to assess parental consistency of discipline completed by parents. Minimum score = 1. Maximum score = 5. High score is better outcome.
Time Frame: 1 month
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Number analyzed (Participants) | 81 | 50
score on a scale | 4.27 (0.14) | 4.05 (0.17)
Statistical Analysis 1: Comparison: Online New Beginnings Program (eNBP) vs Wait-list Control Condition; Test type: Equivalence — Testing the equivalence of the means using two-tailed test; p = 0.01, ANCOVA; Mean Difference (Net) = 0.22, Standard Error of Mean 0.09

8. Primary Outcome: Children's Report of Parent Behavior Inventory -- Consistency Discipline Subscale (Shaefer, 1965) -- Child Report Version
Description: 8-item scales to assess parental consistency of discipline completed by children. Minimum score = 1. Maximum score = 5. High score is better outcome.
Time Frame: 1 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Number analyzed (Participants) | 59 | 43
score on a scale | 4.46 (0.12) | 4.07 (0.16)
Statistical Analysis 1: Comparison: Online New Beginnings Program (eNBP) vs Wait-list Control Condition; Test type: Equivalence — Testing the equivalence of the means using two-tailed test; p = 0.04, ANCOVA; Mean Difference (Net) = 0.38, Standard Error of Mean 0.19

9. Primary Outcome: Oregon Discipline Scale - Follow-Through (Oregon Social Learning Center, 1991) -- Parent Report Version
Description: 11-item scales to assess parental follow-through of discipline completed by parents. Minimum score = 1. Maximum score = 5. High score is better outcome.
Time Frame: 1 month
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Number analyzed (Participants) | 81 | 50
score on a scale | 3.77 (0.16) | 3.55 (0.19)
Statistical Analysis 1: Comparison: Online New Beginnings Program (eNBP) vs Wait-list Control Condition; Test type: Equivalence — Testing the equivalence of the means using two-tailed test; p = 0.02, ANCOVA; Mean Difference (Net) = 0.22, Standard Error of Mean 0.10

10. Primary Outcome: Oregon Discipline Scale - Follow-Through (Oregon Social Learning Center, 1991) -- Child Report Version
Description: 7-item scales to assess parental follow-through of discipline completed by children. Minimum score = 1. Maximum score = 5. High score is better outcome.
Time Frame: 1 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Number analyzed (Participants) | 59 | 43
score on a scale | 4.17 (0.09) | 3.77 (0.10)
Statistical Analysis 1: Comparison: Online New Beginnings Program (eNBP) vs Wait-list Control Condition; Test type: Equivalence — Testing the equivalence of the means using two-tailed test; p = 0.002, ANCOVA; Mean Difference (Net) = 0.40, Standard Error of Mean 0.13

11. Primary Outcome: Child Monitoring Scale (Hetherington et al., 1992) -- Parent Report Version
Description: 9-item scales to assess parental monitoring of child behaviors with friends and at school completed by parents. Minimum score = 1. Maximum score = 5. High score is better outcome.
Time Frame: 1 month
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Number analyzed (Participants) | 81 | 50
score on a scale | 4.71 (0.17) | 4.62 (0.20)
Statistical Analysis 1: Comparison: Online New Beginnings Program (eNBP) vs Wait-list Control Condition; Test type: Equivalence — Testing the equivalence of the means using two-tailed test; p = 0.43, ANCOVA; Mean Difference (Net) = 0.08, Standard Error of Mean 0.10

12. Primary Outcome: Child Monitoring Scale (Hetherington et al., 1992) -- Child Report Version
Description: 9-item scales to assess parental monitoring of child behaviors with friends and at school completed by children. Minimum score = 1. Maximum score = 5. High score is better outcome.
Time Frame: 1 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Number analyzed (Participants) | 59 | 43
score on a scale | 4.45 (0.08) | 4.23 (0.12)
Statistical Analysis 1: Comparison: Online New Beginnings Program (eNBP) vs Wait-list Control Condition; Test type: Equivalence — Testing the equivalence of the means using two-tailed test; p = 0.12, ANCOVA; Mean Difference (Net) = 0.22, Standard Error of Mean 0.14

13. Primary Outcome: Parent Adolescent Communication Scale (Barnes & Olson, 1985) -- Parent Report
Description: 10-item scale to assess parent-child communication completed by parents. Minimum score = 1. Maximum score = 5. High score is better outcome.
Time Frame: 1 month
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Number analyzed (Participants) | 81 | 50
score on a scale | 4.53 (0.13) | 4.36 (0.16)
Statistical Analysis 1: Comparison: Online New Beginnings Program (eNBP) vs Wait-list Control Condition; Test type: Equivalence — Testing the equivalence of the means using two-tailed test; p = 0.03, ANCOVA; Mean Difference (Net) = 0.17, Standard Error of Mean 0.08

14. Primary Outcome: Caught in the Middle Scale (Buchanan et al., 1991) -- Child Report
Description: 7-item scales to assess children being caught in the middle between parents completed by children. Minimum score = 1. Maximum score = 4. High score is worse outcome.
Time Frame: 1 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Number analyzed (Participants) | 59 | 43
score on a scale | 1.49 (0.08) | 1.55 (0.10)
Statistical Analysis 1: Comparison: Online New Beginnings Program (eNBP) vs Wait-list Control Condition; Test type: Equivalence — Testing the equivalence of the means using two-tailed test; p = 0.63, ANCOVA; Mean Difference (Net) = -0.06, Standard Error of Mean 0.13

15. Primary Outcome: Brief Problem Monitor -- Externalizing Subscale (Achenbach et al., 2011) -- Parent Report Version
Description: 7-item scale assessing child externalizing problems as reported by parents. The sum score of the items (range 0-2 for each item) for each individual is converted to T-score, using the algorithm purchased from ASEBA (Achenbach System of Empirically Based Assessment). The range of the T-scores is: 0 (minimum) to 100 (maximum). High score is worse outcome.
Time Frame: 1 month
Measure: Least Squares Mean (Standard Error); unit: T-score on a scale
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Number analyzed (Participants) | 81 | 50
T-score on a scale | 54.72 (1.32) | 55.58 (1.58)
Statistical Analysis 1: Comparison: Online New Beginnings Program (eNBP) vs Wait-list Control Condition; Test type: Equivalence — Testing the equivalence of the means using two-tailed test; p = 0.29, ANCOVA; Mean Difference (Net) = -0.85, Standard Error of Mean 0.80

16. Primary Outcome: Brief Problem Monitor -- Externalizing Subscale (Achenbach et al., 2011) -- Child Report Version
Description: 7-item scale assessing child externalizing problems as reported by children. Item scores range from 0-2, a sum score across the items was computed and converted to a T-score using the algorithm purchased from ASEBA (Achenbach System of Empirically Based Assessment). The range of the T-scores is: 0 (minimum) to 100 (maximum). Score of 50 = the fiftieth percentile of the normative sample. (Achenbach & Rescola, 2001). T-scores of 65 and above are considered sufficiently elevated to be of concern.
  The values shown are the T-score values for the sample. Higher scores indicate a worse outcome.
Time Frame: 1 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: T-score on a scale
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Number analyzed (Participants) | 59 | 43
T-score on a scale | 52.61 (0.66) | 53.68 (0.92)
Statistical Analysis 1: Comparison: Online New Beginnings Program (eNBP) vs Wait-list Control Condition; Test type: Equivalence — Testing the equivalence of the means using two-tailed test; p = 0.33, ANCOVA; Mean Difference (Net) = -1.08, Standard Error of Mean 1.12

17. Primary Outcome: Brief Problem Monitor -- Internalizing Subscale (Achenbach et al., 2011) -- Parent Report Version
Description: 6-item scale assessing child internalizing problems as reported by parents. Item scores range from 0-2, a sum score across the items was computed and converted to a T-score using the algorithm purchased from ASEBA (Achenbach System of Empirically Based Assessment). The range of the T-scores is: 0 (minimum) to 100 (maximum). Score of 50 = the fiftieth percentile of the normative sample. (Achenbach & Rescola, 2001). T-scores of 65 and above are considered sufficiently elevated to be of concern.
  The values shown are the T-score values for the sample. Higher scores indicate a worse outcome..
Time Frame: 1 month
Measure: Least Squares Mean (Standard Error); unit: T-score on a scale
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Number analyzed (Participants) | 81 | 50
T-score on a scale | 56.80 (1.68) | 59.72 (2.00)
Statistical Analysis 1: Comparison: Online New Beginnings Program (eNBP) vs Wait-list Control Condition; Test type: Equivalence — Testing the equivalence of the means using two-tailed test; p = 0.005, ANCOVA; Mean Difference (Net) = -2.92, Standard Error of Mean 1.03

18. Secondary Outcome: Strengths and Difficulties Questionnaire -- Prosocial Subscale (Goodman, 2001) -- Parent Report Version
Description: 5-item scale assessing child prosocial skills as reported by parents. Each of the 5 items is scored 0-2. The score reported is the mean item score. A high score is a better outcome.
Time Frame: 1 month
Measure: Least Squares Mean (Standard Error); unit: Sum score on a scale
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Number analyzed (Participants) | 81 | 50
Sum score on a scale | 1.65 (0.11) | 1.59 (0.13)
Statistical Analysis 1: Comparison: Online New Beginnings Program (eNBP) vs Wait-list Control Condition; Test type: Equivalence — Testing the equivalence of the means using two-tailed test; p = 0.42, ANCOVA; Mean Difference (Net) = 0.07, Standard Error of Mean 0.08

19. Secondary Outcome: Strengths and Difficulties Questionnaire -- Prosocial Subscale (Goodman, 2001) -- Child Report Version
Description: Each of the 5 items is scored 0-2 (range 0-10). The score reported is the mean of the total scores. A higher score is a better outcome.
Time Frame: 1 month
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Sum score on a scale
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
Number analyzed (Participants) | 59 | 43
Sum score on a scale | 8.90 (0.20) | 8.89 (0.24)
Statistical Analysis 1: Comparison: Online New Beginnings Program (eNBP) vs Wait-list Control Condition; Test type: Equivalence — Testing the equivalence of the means using two-tailed test; p = 0.97, ANCOVA; Mean Difference (Net) = 0.01, Standard Error of Mean 0.30

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the full course of the trial, 12 weeks.
Description: No adverse events occurred from baseline through post test.
Arm/Group | Online New Beginnings Program (eNBP) | Wait-list Control Condition
All-Cause Mortality (participants affected / at risk) | 0/140 | 0/93
Serious Adverse Events (participants affected / at risk) | 0/140 | 0/93
Other Adverse Events (participants affected / at risk) | 0/140 | 0/93

LIMITATIONS AND CAVEATS:
Limitations are that only pre and post assessment was completed with no follow-up over time.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-27): https://cdn.clinicaltrials.gov/large-docs/32/NCT05209932/Prot_SAP_001.pdf